CLINICAL TRIAL: NCT01041690
Title: Bevacizumab (Avastin) as an Adjunct to Vitrectomy in the Management of Severe Proliferative Diabetic Retinopathy: a Prospective Case Series
Brief Title: Efficacy of PreOperative Bevacizumab for Diabetic Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Tamer Ahmed Macky, Cairo University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Beva-Cairo-A1
Record Dates: First submitted 2009-12-31; First posted 2010-01-01 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2007-01

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative Diabetic Retinopathy; Vitrectomy; Bevacizumab
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
Reports of the use of intravitreal bevacizumab (Avastin, Genentech) for the reduction of neovascularization in proliferative diabetic retinopathy have demonstrated significant regression in the number of new vessels. Reducing the vascularity of neovascular fibrovascular tissue can potentially reduce bleeding intraoperatively and thus facilitate the vitrectomy procedure. The investigators chose to investigate the potential benefit of the use of preoperative bevacizumab in the management of these most complex cases.

DETAILED DESCRIPTION:
PURPOSE: To evaluate the role of preoperative intravitreal bevacizumab as an adjunct to vitrectomy in the management of severe diabetic eye disease.

SETTINGS: Kasr El-Aini Teaching Hospital - Cairo University from 2007 to 2008. METHODS: Twenty eyes of 19 patients with severe proliferative diabetic retinopathy were recruited into the study. All eyes underwent a single intravitreal injection of bevacizumab 1.25 mg in 0.05 ml one week prior to vitrectomy for tractional (14), combined tractional/rhegmatogenous retinal detachment (4), and fibrovascular tissue covering/distorting the macula (2). Exclusion criteria were: previous vitrectomy, neovascular glaucoma, and dense media opacity (dense cataract and vitreous hemorrhage) precluding fluorescein angiography (FA) that was done pre- and 1 week post injections. Best corrected visual acuity (BCVA), anterior segment with dilated fundus examinations, and intraocular pressures (IOP), were done pre-, 1 week post-injections, 1 day, 1 week and monthly for 3 months post-vitrectomy. Intra- and post-operative bleedings were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Tractional Retinal Detachment involving or threatening the macula,
* Tractional+Rhegmatogenous Retinal Detachment, or
* Fibrovascular tissue covering and distorting the macula.

Exclusion Criteria:

* Vitrectomy
* Neovascular glaucoma
* Dense media opacity (dense cataract and vitreous hemorrhage) precluding fluorescein angiography (FA)

Ages: 9 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Intra- and post-operative bleedings were recorded. | 3 months

SECONDARY OUTCOMES:
Best Corrected Visual Acuity | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department Of Ophthalmology, Cairo, Cairo Governorate, Egypt